CLINICAL TRIAL: NCT05869110
Title: OLFO-FOOD: OLFactory Odour Stimulation and FOOD Preferences
Brief Title: OLFactory Odour Stimulation and FOOD Preferences
Acronym: OLFO-FOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-00511, kt23Timper
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: olfactory stimulation; Hunger; Appetite; calorie intake; food choice; metabolic parameters
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, single-blind, cross-over, single-centre trial
Who Masked: Participant
Masking Description: Study participants will not be informed which substances are investigated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (Experimental): Olfactory stimulation
  Interventions: Other: Effects of odours on calorie intake, food choice and metabolic parameters
- Placebo (Placebo Comparator): Propylene glycol
  Interventions: Other: Effects of odours on calorie intake, food choice and metabolic parameters

INTERVENTIONS:
Other: Effects of odours on calorie intake, food choice and metabolic parameters — Evaluation of the effects of olfactory stimulation compared to placebo on calorie intake and preference of food during a test-buffet.
  Odours will be assigned in a randomized order. Each participant will receive both odours, in between there will be a wash-out period of 1 week.

SUMMARY:
The aim of the present "OLFO-FOOD" clinical trial is to investigate, if olfactory stimulation impacts food choice, reference and calorie intake in humans with obesity assessed using a test buffet.

DETAILED DESCRIPTION:
Overweight study participants will be included in this study. For the participants the study consists of the screening visit and main visit 1 and 2. In between the main visits there is a wash-out period of 1 week (7 days ± 3 days). In total, participants will have 3 visits. After the screening visit and before the main visit 1, odours will be assigned in a randomized order. Each participant will receive both odours. The two visits (main visit 1 and 2) will have the exact same procedures except for the olfactory odour.

Hunger, appetite, thirst, food perception, nausea, headache and mood will be assessed and the first blood samples will be collected. The participants will receive the aspUraclip® filled with 50 μl of either olfactory stimulation or placebo (propylene glycol), due to the computer-generated randomization order. The "aspUraclip®" will be clipped to the nasal septum for 15 minutes. After olfactory stimulation, vital parameters will be measured and blood samples will be taken. Participants will rate hunger, appetite, thirst, nausea, headache, mood, as well as local nose irritation, odour intensity and odour perception. Directly afterwards, the participants choose food ad libitum from a test-buffet. Participants will have 2 hours to eat from the buffet, but can finish earlier if they wish. Eating time will be recorded. After finishing their meal, vitals will be measured, blood samples will be collected and the participants will rate hunger, appetite (general, carbohydrates, meat, dairy foods, vegetables, fruits, sweets, salty foods), thirst, nausea, headache, mood, food taste, food taste intensity, food scent intensity and food scent perception on a 10-point VAS (visual analogue scale). 2 hours after the start of the test-buffet, patients will rate the same questions on a VAS again, vitals and blood samples will be taken. If the participants eat throughout the 2-hour-timespan of the test-buffet and don't stop early, there will be only one measurement (vitals, VAS, BS) after 2 hours, when the test-buffet ends. Food intake will be measured by weighing the food before and after consumption. Following the test-buffet, patients will have a resting phase of 2 hours. During this phase, patients are free to read, listen to music or similar. After the 2 hour resting phase, vitals will be measured, blood samples collected and VAS-questions asked.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Written informed consent
* BMI ≥30 kg/m2
* Normosmia (as defined by Sniffin' Sticks Test)

Exclusion Criteria:

* Known allergy to olfactory stimulation substance, citrus fruits, citrus flavours, citrus food products
* Lactose-intolerance, celiac disease or non-celiac wheat sensitivity
* Diet other than omnivore or vegetarian
* Eating disorder (now or in the past)
* Dysphagia
* Acute disease affecting food intake
* Acute upper respiratory tract infection, acute or chronic sinusitis
* Severe visual impairment (vision <10%)
* Surgical intervention of the nasal cavity or the paranasal sinus
* Current illicit drug abuse including daily marijuana and CBD (Cannabidiol) consumption (alcohol ≤2 drinks per day allowed)
* Any kind of severe chronic disease (e.g. severe heart failure, active cancer disease)
* Type 1 and 2 diabetes mellitus
* Treatment with insulin-sensitizing drugs within the last 3 months
* Treatment with Glucagon-like Peptide 1 (GLP1)-analoga
* History of neurodegenerative diseases, severe head trauma
* Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2)
* Known liver cirrhosis or other severe liver impairment
* Use of any kind of decongestant more than twice a week
* Uncontrolled dysthyroidism
* Uncontrolled hypertension
* Regular use of psychopharmaceutic drugs
* Study participants aims to start a new diet or exercise program during the study
* Bariatric surgery
* Pregnancy/Lactation
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in an interventional study within the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Change in calorie intake after olfactory stimulation | two time assessment at baseline and after 1 week
  Olfactory stimulation compared to placebo in participants with obesity with a BMI ≥30 kg/m2 assessed by a test-buffet.

SECONDARY OUTCOMES:
Change in food preference after olfactory stimulation | two time assessment at baseline and after 1 week
  Olfactory stimulation compared to placebo in participants with obesity with a BMI ≥30 kg/m2 assessed by a test-buffet.
  Proportion of carbohydrates, fat and protein of the chosen food products (processed foods, warmed-up ready-to-eat meal, fresh fruits and vegetables)
Change of hunger assessed via VAS (Visual Analogue Scale) upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Hunger will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change of appetite assessed via (Visual Analogue Scale) VAS upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Appetite will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change of thirst assessed via (Visual Analogue Scale) VAS upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Thirst will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change of nausea assessed via (Visual Analogue Scale) VAS upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Nausea will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change of headache assessed via (Visual Analogue Scale) VAS upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Headache will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change of mood assessed via (Visual Analogue Scale) VAS upon olfactory stimulation | up to eight time assessment from baseline till day 7
  Mood will be assessed via 10-point VAS Score (0= not at all, 10= maximum)) upon olfactory stimulation compared to placebo before and directly after olfactory stimulation, before and after exposure to a test-buffet.
Change in plasma glucose Level (mmol/L) | up to 10 time assessment at visit one (Baseline, TB0, TBX, TB2, TBR) and after 1 week at visit 2 (Baseline TB0, TBX, TB2, TBR)
  Up to 5 blood samplings will be collected during each main visit, depending on the individual endpoint at the test-buffet: 4 blood samplings (60.8ml) if the participant eats the full 2 hours from the test-buffet, 5 samplings (76ml) if the participant stops eating from the test-buffet early.
  * Before olfactory stimulation (OS), (Baseline)
  * After OS, before the test-buffet (TB0)
  * After individual endpoint at the test-buffet (TBX)
  * After 2 hours of test-buffet (TB2)
  * After 2 hours of resting phase (TBR)
Change in plasma insulin Level (pmol/L) | up to 10 time assessment at visit one (Baseline, TB0, TBX, TB2, TBR) and after 1 week at visit 2 (Baseline TB0, TBX, TB2, TBR)
  Up to 5 blood samplings will be collected during each main visit, depending on the individual endpoint at the test-buffet: 4 blood samplings (60.8ml) if the participant eats the full 2 hours from the test-buffet, 5 samplings (76ml) if the participant stops eating from the test-buffet early.
  * Before OS (Baseline)
  * After OS, before the test-buffet (TB0)
  * After individual endpoint at the test-buffet (TBX)
  * After 2 hours of test-buffet (TB2)
  * After 2 hours of resting phase (TBR)
Change in serum cortisol Level (nmol/L) | up to 10 time assessment at visit one (Baseline, TB0, TBX, TB2, TBR) and after 1 week at visit 2 (Baseline TB0, TBX, TB2, TBR)
  Up to 5 blood samplings will be collected during each main visit, depending on the individual endpoint at the test-buffet: 4 blood samplings (60.8ml) if the participant eats the full 2 hours from the test-buffet, 5 samplings (76ml) if the participant stops eating from the test-buffet early.
  * Before OS (Baseline)
  * After OS, before the test-buffet (TB0)
  * After individual endpoint at the test-buffet (TBX)
  * After 2 hours of test-buffet (TB2)
  * After 2 hours of resting phase (TBR)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Timper, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland